CLINICAL TRIAL: NCT03692065
Title: Long-term Treatment of Cancer Associated VTE: Reduced vs Full Dose of Apixaban : API-CAT STUDY for APIxaban Cancer Associated Thrombosis
Brief Title: API-CAT STUDY for APIxaban Cancer Associated Thrombosis
Acronym: API-CAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P170604J
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Cancer-associated Thrombosis
Keywords: Cancer; VTE; Apixaban; Thrombosis
MeSH Terms: conditions — Neoplasms; Thrombosis | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban film coated tablets 2.5 mg (Active Comparator): Patients randomized in the apixaban reduced dose group will receive an apixaban 2.5 mg tablet and a placebo of apixaban 5 mg tablet, twice daily for 12 months.
  Interventions: Drug: Apixaban 5 MG
- Apixaban film coated tablets 5 mg (Active Comparator): Patients randomized in the apixaban full dose group will receive a placebo of apixaban 2.5 mg tablet and an apixaban 5 mg tablet, twice daily for 12 months.
  Interventions: Drug: Apixaban 5 MG

INTERVENTIONS:
Drug: Apixaban 5 MG — Subjects will be randomized (1:1 ratio) to apixaban 5 mg bid (full dose) or apixaban 2.5 mg bid (reduced-dose) using a centralized IWRS (double blind study).
  Other Names: Apixaban 2.5 MG

SUMMARY:
The main objective is to determine whether a low-dose regimen of apixaban (2.5 mg bid) is non inferior to a full-dose regimen of apixaban (5 mg bid) for the prevention of recurrent venous thromboembolism (VTE) in patients with active cancer who have completed at least 6 months of anticoagulant therapy for treating a documented index event of proximal deep venous thrombosis (DVT) (symptomatic or incidental) or pulmonary embolism (symptomatic or incidental).

DETAILED DESCRIPTION:
For patients completing at least 6 months of anticoagulant therapy in whom the cancer is active, the thrombotic risk is arguably ongoing and indefinite anticoagulation seems required.

Given apixaban 5 mg bid is an alternative for the first 6 months of treatment, we intend to assess whether it is possible to lower the dose of apixaban (2.5 mg bid) after completing at least 6 months of anticoagulant treatment in a specific population of patients with cancer associated thrombosis (CAT) requiring extended anticoagulant treatment and with significant life expectancy. There are 2 conditions to be met : demonstrate the non-inferiority of the 2.5 mg bid regimen on the efficacy endpoint and then demonstrate the superiority of the 2.5 mg bid regimen as compared to the 5 mg bid on the safety endpoint.

It is a multicenter, international, prospective, randomized, parallel-group, double-blind non-inferiority trial with blinded adjudication of outcome events (approximately 160 centers in approximately 10 countries (France, Italy, Spain, Belgium, Greece, Netherlands, UK, Switzerland, Poland, Austria), with a number of expected inclusions of 11 patients per site.

Subjects should be randomized within 7 days after the last dose of their initial 6-month treatment, defined as the treatment ongoing after completing at least 6 months of anticoagulant treatment from the beginning of the anticoagulant treatment for the index event. This treatment may be low-molecular weight heparin (LMWH), direct oral anticoagulant (DOAC) or vitamin K antagonist (VKA). If a VKA was used as standard anticoagulant therapy, then an INR must be documented as 2 or less before randomization. Every attempt should be made to randomize subjects as soon as possible after the initial treatment has been discontinued.

Subjects will be stratified based on the cancer site and the type of disease treated (PE with/without DVT or DVT alone). If a subject had both symptomatic DVT and symptomatic PE, the subject will be stratified as having symptomatic PE.

ELIGIBILITY:
Minimum Age: 18 Years

Maximum Age:

Sex: All Gender Based: No Accepts Healthy Volunteers: No

Criteria:

Inclusion Criteria:

* Signed written informed consent
* Any cancer diagnosed histologically (other than basal-cell or squamous-cell carcinoma of the skin, primary brain tumor or intra-cerebral metastasis)
* Active cancer defined as the presence of measurable disease or ongoing (or planned) chemotherapy, radiotherapy, hormonotherapy, targeted therapy, immunotherapy at inclusion
* Objectively documented index event : Symptomatic or incidental proximal lower-limb, iliac, inferior vena cava DVT or symptomatic or incidental pulmonary embolism in a segmental or larger pulmonary artery or incidental PE in a segmental or larger pulmonary artery

  1. Proximal DVT is defined as DVT that involves at least the popliteal vein or a more proximal vein, demonstrated by imaging with compression ultrasound (CUS), including grey-scale or color-coded Doppler, or ascending contrast venography or contrast enhanced computed tomography or magnetic resonance imaging
  2. PE has to be demonstrated by imaging as follows:

     * an intraluminal filling defect in segmental or more proximal branches on contrast enhanced chest computed tomography or on computed tomography pulmonary angiography; or
     * an intraluminal filling defect or a sudden cutoff of vessels more than 2.5 mm in diameter on the pulmonary angiogram; or
     * a perfusion defect of at least 75% of a segment with a local normal ventilation result (high-probability) on ventilation/perfusion lung scan (VPLS)
  3. Incidental VTE is defined as proximal DVT or PE detected by imaging incidentally when a patient undergoes imaging studies as standard of care for the management of his or her malignancy or other reasons but not for a VTE suspicion(e.g. cancer diagnosis or staging).
* Completed at least 6 months of anticoagulant therapy at therapeutic dosage (whatever the drug and the dosing),or completed assigned a clinical trial study treatment, for the treatment of the index event and patient still receiving anticoagulant treatment 6 months after occurrence of the VTE index
* No objectively documented symptomatic recurrence of VTE between the index event and randomization.
* Anticipated duration of anticoagulant treatment of at least 12 months at the time of randomization
* Patient affiliated to social security for French centers.

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method of birth control [such as oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (condoms)] to avoid pregnancy for the entire study
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or prior to investigational product administration
* Isolated sub-segmental (incidental or symptomatic) PE without associated DVT
* Isolated distal DVT of the legs
* Isolated upper-extremity DVT or superior vena cava thrombosis
* Isolated visceral thrombosis
* Isolated catheter thrombosis
* Objectively documented symptomatic recurrence of VTE after the index event under anticoagulant treatment
* VTE during anticoagulant treatment given at therapeutic dosage
* Subjects with indications for long-term treatment with a VKA, such as:
* Mechanical heart valve
* Antiphospholipid syndrome
* Subjects with indication for long-term anticoagulation with a VKA or a DOAC at therapeutic dosage
* Conditions increasing the risk of serious bleeding

  1. intracranial or intraocular bleeding within the 6 months
  2. major surgery within 2 weeks prior to randomization
  3. overt major bleeding at time of randomization
* Life expectancy < 12 months
* Eastern Cooperative Oncology Group (ECOG) level 3 or 4
* Bacterial endocarditis
* Uncontrolled hypertension: systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg
* Platelet count < 75,000/mm3
* Hemoglobin < 8g /dl
* Creatinine clearance < 30 ml /min based on the Cockcroft Gault equation
* Acute hepatitis, chronic active hepatitis, liver cirrhosis; or an alanine aminotransferase level 3 times or more and/or bilirubin level 2 times or more higher the upper limit of the normal range
* Subjects requiring acetylsalicylic acid >165 mg/day at randomization or thienopyridine therapy (clopidogrel, prasugrel, or ticagrelor).
* Subjects requiring dual anti-platelet therapy (such as acetylsalicylic acid plus clopidogrel or acetylsalicylic acid plus ticlopidine) at randomization. Subjects who transition from dual antiplatelet therapy to monotherapy prior to randomization will be eligible for the trial.
* Concomitant use of strong inhibitors of both cytochrome P-450 3A4 and P Glycoprotein (e.g., human immunodeficiency virus protease inhibitors or systemic ketoconazole) or strong inducers of both cytochrome P450 3A4 and P Glycoprotein (e.g.,rifampicin, carbamazepine, or phenytoin).
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
* Hypersensitivity to apixaban
* Subjects participating in another pharmaco therapeutic program with an experimental therapy that is known to affect the coagulation system
* Under 18 years old
* Patients under legal protection (guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1766 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
The incidence of an an adjudicated composite endpoint | During the treatment period (12 months)
  The incidence of an adjudicated composite of recurrent symptomatic VTE (proximal and/or distal DVT and/or symptomatic PE and/or upper limb or central venous catheter thrombosis or incidental VTE (proximal DVT or PE), or death due to PE during the treatment period.
  Incidental VTE is defined as proximal DVT or PE detected by imaging incidentally when a patient undergoes imaging studies as standard of care for the management of the malignancy or other reasons but not for a VTE suspicion.

SECONDARY OUTCOMES:
The incidence of adjudicated major and clinically relevant non-major bleeding | During the treatment period (12 months)
  The definition of major bleeding described is adapted from the International Society on Thrombosis and Hemostasis (ISTH) definition (Schulman JTH 2005).
Recurrent symptomatic VTE | During the treatment period (12 months)
  Recurrent VTE objectively confirmed after clinical suspicion
VTE related-death | During the treatment period (12 months)
  VTE related-death: PE based on objective diagnostic testing, autopsy, or sudden death; i.e. death occurring within one hour of the onset of new symptoms which cannot be attributed to a documented cause (unexplained death) and for which PE/DVT cannot be ruled out as the cause.
All-cause death | During the treatment period (12 months)
  All deaths will be adjudicated by the ICAC and classified as either VTE-related, cancer death (including all deaths due to the underlying cancer), bleeding-related or others, including all deaths due to a clearly documented other cause, such as respiratory failure (e.g., terminal emphysema), infections/sepsis etc.
Adjudicated major bleeding. | During the treatment period (12 months)
  The definition of major bleeding described is adapted from the International Society on Thrombosis and Hemostasis (ISTH) definition (Schulman 2005) and includes
  * Acute clinically overt bleeding with one or more of the following:
    * A decrease in hemoglobin (Hgb) of 2 g/dL or more
    * A transfusion of 2 or more units of packed red blood cells
    * Symptomatic bleeding that occurs in at least one of the following critical sites:
      * Intracranial
      * Intraspinal
      * Intraocular (within the corpus of the eye; thus, a conjunctival bleed is not an intraocular bleed)
      * Pericardial
      * Intra-articular
      * Intramuscular with compartment syndrome
      * Retroperitoneal
  * Bleeding that is fatal: bleeding event that the independent adjudication committee determines is the primary cause of death or contributes directly to death.
Adjudicated composite of recurrent symptomatic VTE, VTE related-death, all-cause death, adjudicated major bleeding. | During the treatment period (12 months)
  Adjudicated composite of recurrent symptomatic VTE, VTE related-death, all-cause death, adjudicated major bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Meyer, Pr, Study Director — APHP(ASSISTANCE PUBLIQUE DES HOPITAUX DE PARIS
Locations (114):
- Austria (4):
  - Medical university of Graz, Graz
  - Medical university of Innsbruck, Innsbruck
  - Ordensklinikum Linz gmbH Elisabethinen, Linz
  - Medical university of Vienna, Vienna
- Belgium (7):
  - Erasmus Hospital Brussel, Brussels
  - Institut Roi Albert II, Brussels
  - AZ Groeninge, Kortrijk
  - Uz Leuven, Leuven
  - CHC Saint-Joseph, Liège
  - CHR de la Citadelle, Liège
  - CHU de Liège, Liège
- Canada (5):
  - University of Calgary, Calgary
  - University of Alberta, Edmonton
  - Ottawa Hospital Research Institute OTTAWA, Ottawa
  - Toronto General Hospital, Toronto
  - Diamond Health Care Centre, Vancouver
- France (68):
  - C.H.U. D'Amiens Picardie, Amiens
  - Chu D'Angers, Angers
  - HÔPITAL PRIVÉ ARRAS LES BONNETTES - Espace Artois Santé, Arras
  - Centre Hospitalier d'Avignon, Avignon
  - Institut Sainte Catherine, Avignon
  - Hopital Jean Minjoz, Besançon
  - Hôpital AVICENNE - APHP, Bobigny
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Hôpital d'Instruction des Armées Clermont Tonnerre, Brest
  - Chru Brest - Hopital Morvan, Brest
  - Chru Brest- Hopital Cavale Blanche, Brest
  - Centre François Baclesse, Caen
  - Centre de Recherche Clinique, Caen
  - Hopital Cote de Nacre, Caen
  - Clinique Du Parc, Castelnau-le-Lez
  - Centre hospitalier Métropole Savoie, Chambéry
  - Ch Cholet, Cholet
  - Hia Percy, Clamart
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hôpital BEAUJON - APHP, Clichy
  - Hôpital Henri Mondor, Créteil
  - Hôpital HENRI MONDOR - APHP, Créteil
  - CHU DIJON BOURGOGNE - Hôpital François Mitterrand, Dijon
  - Chu de Grenoble, Grenoble
  - Chd Vendee, La Roche-sur-Yon
  - Centre Hospitalier Du Mans, Le Mans
  - Centre hospitalier Emile Roux, Le Puy-en-Velay
  - Chu de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Hôpital Prive Jean Mermoz, Lyon
  - Clinique de l'Infirmerie Protestante de Lyon, Lyon
  - Hopital La Timone Adultes, Marseille
  - Groupe hospitalier sud Ile de France, Melun
  - Hopital Saint- Eloi, Montpellier
  - C.H. Des Pays de Morlaix, Morlaix
  - Centre D Oncologie de Gentilly, Nancy
  - CHU DE Nantes - Site Hotel Dieu, Nantes
  - Chu de Nice, Nice
  - Institut Curie, Paris
  - Hôpital Saint Antoine - APHP, Paris
  - Hôpital PITIE SALPETRIERE - APHP, Paris
  - Hôpital COCHIN - APHP, Paris
  - Hôpital GEORGES POMPIDOU - APHP, Paris
  - Hôpital Bichat Claude Bernard, Paris
  - Hopital Tenon - Aphp, Paris
  - Hopital Saint-Joseph, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Polyclinique de Courlancy, Reims
  - CHU de Rennes, Rennes
  - Centre Anti-Cancereux E. Marquis, Rennes
  - Chu de Rouen - Hopital Charles Nicolle, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Hôpital Nord, Saint-Etienne
  - C.H.I Poissy-Saint Germain, Saint-Germain-en-Laye
  - Centre Hospitalier de Saint Malo, St-Malo
  - Clinique de l' Estrée, Stains
  - Clinique Saint Anne, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Hopital Foch, Suresnes
  - Chi de Toulon La Seyne, Toulon
  - Iuct Oncopole, Toulouse
  - Hopital Andre Mignot, Versailles
  - L'Hôpital Nord-Ouest, Villefranche-sur-Saône
  - Hôpital Paul Brousse - APHP, Villejuif
  - Institut Gustave Roussy, Villejuif
  - Médipôle Hôpital Mutualiste, Villeurbanne
  - Hopital Louis Mourier - APHP, Colombes, Île-de-France Region
- Greece (4):
  - Athens School of Medicine, Athens
  - National and Kapodistrian University of Athens ALEXANDRA Hospital, Athens
  - University General Hospital "Attikon", Athens
  - University of Athens, Athens
- Italy (3):
  - Ospedale di Castelfranco Veneto, Castelfranco Veneto
  - Opedale clinicizzato colle dell'ara, Chieti
  - Universita di Perugia, Perugia
- Netherlands (7):
  - Amsterdam university medical center, Amsterdam
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - Rode Kruis Ziekenhuis, Beverwijk
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Tergooi Hospital Hilversum, Hilversum
  - Leiden university medical center, Leiden
  - Diakonessenhuis, Utrecht
- Centre of postgraduate medical education at the european health centre Otwock, Otwock, Poland
- Spain (11):
  - Hospital genarl Univ de Albacete, Albacete
  - Hospital Virgen de los lirios, Alicante
  - Fundacio Hospital de L'Esperit Sant, Barcelona
  - Hospital universitari Germans trias i Pujol, Barcelona
  - Parc Santari Sant Joan de Deu - Hospital general, Barcelona
  - Hospital general Universitario Santa Lucia, Cartagena
  - Hospital general universitario de ciudad real, Ciudad Real
  - Hospital Olot i Comarcal de ma Garrotxa, Girona
  - Hospital universitari de Girona, Girona
  - Hospital universitario Infanta Sofia, Madrid
  - Hospital universitario Virgen del Rocio, Seville
- Switzerland (3):
  - Istituto Oncologico della svizzera Italiana, Bellinzona
  - Hopitaux universitaires de Genève, Geneva
  - Lausanne university hospital - CHUV, Lausanne
- Queens centre castle hill hospital, Cottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahe I, Chapelle C, Girard P, Carrier M, Palomares LJ, Samama CM, Helfer H, Gerotziafas G, Laporte S, Vicaut E, Mismetti P; API-CAT Study Group; API-CAT Investigators. Predictors of clinically relevant bleeding during extended anticoagulation for cancer-associated venous thromboembolism (API-CAT): a post-hoc analysis of a randomised, non-inferiority trial. Lancet Haematol. 2026 Jan;13(1):e41-e48. doi: 10.1016/S2352-3026(25)00291-1. Epub 2025 Dec 6. PMID 41365312
- [Derived] Mahe I, Carrier M, Mayeur D, Chidiac J, Vicaut E, Falvo N, Sanchez O, Grange C, Monreal M, Lopez-Nunez JJ, Otero-Candelera R, Le Gal G, Yeo E, Righini M, Robert-Ebadi H, Huisman MV, Klok FA, Westerweel P, Agnelli G, Becattini C, Bamias A, Syrigos K, Szmit S, Torbicki A, Verhamme P, Maraveyas A, Cohen AT, Ay C, Chapelle C, Meyer G, Couturaud F, Mismetti P, Girard P, Bertoletti L, Laporte S; API-CAT Investigators. Extended Reduced-Dose Apixaban for Cancer-Associated Venous Thromboembolism. N Engl J Med. 2025 Apr 10;392(14):1363-1373. doi: 10.1056/NEJMoa2416112. Epub 2025 Mar 29. PMID 40162636